CLINICAL TRIAL: NCT06338644
Title: Palbociclib in Metastatic Breast Cancer: Gene Polymorphism-based Study in Egyptian Patients.
Acronym: Palbociclib
Status: Not yet recruiting | Type: Observational
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Yassmin Genina, Assistant lecturer at Faculty of Pharmacy, Helwan University
Other Study IDs: HelwanUY
Record Dates: First submitted 2024-03-24; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Hormone-receptor-positive Breast Cancer; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; Metastatic Breast Cancer
Keywords: Metastatic breast Cancer, Palbociclib, Pharmacogenomic
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Primary resistant to endocrine therapy: Primary endocrine resistance is defined as a relapse within 2 years of adjuvant endocrine treatment or disease progression during the first 6 months of first-line endocrine therapy for advanced or MBC
  Interventions: Drug: Palbociclib
- Secondary resistant to endocrine therapy: Secondary resistance is defined in early BC as a relapse that occurs after at least 2 years of endocrine therapy and during or within the first year of completing adjuvant endocrine therapy. In advanced BC or MBC, secondary resistance is defined as disease progression after more than 6 months of endocrine therapy
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — 3 weeks on, 1 week off

SUMMARY:
Cyclin-dependent kinase (CDK) 4/6 inhibitors are a class of agents recently introduced in the clinic for the treatment of advanced hormone receptor-positive (HR+) and HER2-negative (HER2-) BC. Palbociclib, ribociclib and abemaciclib have all been approved by the US Food and Drug Administration (FDA) and the European Medicines Agency among other regulatory bodies

DETAILED DESCRIPTION:
Several factors are thought to influence the variability of treatment efficacy and toxicity, including organ function, comedications, hormonal status, body weight, age, comorbidities, etc. Among them, single nucleotide polymorphisms (SNPs) as rs1128503, rs2032583 are attracting huge interest to address the interindividual variability in drug response, whether in terms of efficacy or safety

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients (≥18 years). 2. Confirmed diagnosis with MBC. 3. HR-positive/HER2-negative MBC as ascertained by immunohistochemistry (IHC) or fluorescence in situ hybridization in primary or metastatic tissue samples.

  4. Patients with primary or secondary resistance to endocrine therapy. 5. Patients with Eastern Cooperative Oncology Group (ECOG) 0 or 1. 6. Scheduled to receive Palbociclib in first- or second-line metastatic setting.

Exclusion Criteria:

1. Prior exposure to fulvestrant or everolimus.
2. Patients with uncontrolled brain metastases or symptomatic visceral spread who are at risk of life-threatening complications.
3. Patients refusing to sign the written informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hormone receptor-positive HER2-negative metastatic breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
1-year Progression free survival (PFS) | 1 year
  the time from enrollment until first evidence of disease progression or death

SECONDARY OUTCOMES:
Neutropenia | 1 year
  Grade 3 or 4 neutropenia

REFERENCES:
- [Derived] Mohamed Ebid AI, Fahim Genina YM, Shawky Haffez HR, Ahmed Hakam SH, Hassan Kassem LM, Mohamed AbdelMotaleb SM. Palbociclib in endocrine-resistant metastatic breast cancer: real-world outcomes. Expert Rev Anticancer Ther. 2025 Sep 21:1-10. doi: 10.1080/14737140.2025.2560941. Online ahead of print. PMID 40957562